CLINICAL TRIAL: NCT01996124
Title: Acute Effect of Pulmonary Desufflation on Cardiac Performance in COPD Patients in Stable Conditions. Pilot Study
Brief Title: Acute Effect of Pulmonary Desufflation on Cardiac Performance in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Pierachille Santus, Head of Pulmonary Rehabilitation Unit, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 902 CEC
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: COPD; Hyperinflation; Right Cardiac Failure
Keywords: COPD; Pulmonary Hyperinflation; Ultra Long Acting Beta 2 Agonists; Cor Pulmonale; Cardiac performance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Heart Disease | interventions — Fructose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indacaterol (Experimental): Indacaterol Fumarate 150 mcg Breezehaler,Onbrez Novartis International AG, Basel Switzerland. Once daily.
  Interventions: Drug: Indacaterol Fumarate
- Placebo (Placebo Comparator): Placebo Breezehaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol Fumarate — 150 mcg inhalation powder, hard capsules, once daily
  Other Names: Onbrez Breezhaler (Novartis International AG, Basel Switzerland)
  Arms: Indacaterol
Drug: Placebo — Fructose, dry inhalation powder, hard capsules via breezhaler
  Other Names: Placebo, fructose 150 mcg via Breezhaler, inhalation powder
  Arms: Placebo

SUMMARY:
Chronic Obstructive Pulmonary disease (COPD) is one of the major clinical entities that causes thousands of deaths every year all over the world and weights a lot on the health care system of every country in terms of direct and indirect costs. The physiopathological modifications that characterise COPD are represented by irreversible (sometimes partially reversible) airflow obstruction, and bronchiolar inflammation. Lungs that develop emphysema lack of elastic recoil and imply increased resistances and airflow obstruction due to loss of lung parenchyma and supporting elastic structures. All these modifications produce air trapping and so lung hyperinflation. The latter is precisely the cause of the symptoms and particularly dyspnoea which is often heavily perceived by COPD patients and that drives to the limitation of daily activities. Lung hyperinflation and the other alterations that occur in COPD imply gas retention and increase in pulmonary vascular resistances. Considering that the rib cage has limited elastic properties, the effects of gas trapping and lung parenchymal damage on mediastinum and particularly on heart mechanics is indisputable. Together with alveolar hypoxia, lung hyperinflation is responsible for the development, as the disease progresses, of the cor pulmonale. Tha latter causes pulmonary hypertension and increased mechanic load during right heart chambers contraction and relaxation. Those alterations may effect left heart chambers too.

Airflow obstruction in COPD is usually treated by inhaled bronchodilators and corticosteroids. The main and most used bronchodilators are represented by beta 2 agonists (short, long and ultra-long acting) and anticholinergic inhalatory drugs, which can be also short, long and ultra long acting. Among ultra long acting beta 2 agonists, indacaterol is characterised by quick onset of action (5 minutes), and guarantees an effective bronchodilation duration of 24 hours. It is also known that it has an important effect on reducing lung hyperinflation decreasing residual volume and consequently allowing an increase of inspiratory capacity. The purpose of our study is to evaluate the effects of indacaterol on lung hyperinflation in COPD subjects of any stage and with lung air trapping, and the consequent potential effects on heart performance evaluated by cardiac trans thoracic echo color doppler.

DETAILED DESCRIPTION:
In a paper recently published, Barr et al, supposed that pulmonary emphysema and bronchial obstruction were inversely related with ventricular telediastolic volume, with the ejection volume and the ejection fraction in patients with severe pulmonary disease. The mechanisms that are involved in the development of cor pulmonale are the increase of pulmonary vascular resistances, lung hyperinflation and hypoxic vascular constriction. All the mentioned contribute to the generation of right cardiac failure and consequently, left cardiac failure. The authors assessed lung hyperinflation by CT scan, pulmonary function by spirometry, and cardiac kinetic and mechanics by magnetic resonance. They concluded that the amount of emphysema and bronchial obstruction were related with a worse telediastolic left ventricular volume and stroke volume, no relation was found with ejection fraction. It was evident that patients with severe pulmonary disease and with no present cardiac diseases, had sub-clinic modifications that one day may lead them to the development of cor pulmonale.

The effect of bronchodilation, with its effect on lung hyperinflation, may have a role in producing some modifications in this context. That's why that the aim of our study is centered on the evaluation of the effect of bronchodilation firstly on diastolic right ventricular function and also on interventricular septum motility, on the ejection fraction and on the kinetics of right cardiac chambers assessed by cardiac echocardiography

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* COPD patients with age raging from 50 to 85 years old
* Patients with at least a history of COPD of one year
* COPD patients clinically stable in the last three months
* COPD subjects with FEV1 (Forced Expiratory Volume at one second)<70% of predicted value
* FEV1/FVC (Forced Vital Capacity)<88% (males) or <89% (females) of LLN (Lower Levels of Normality)
* COPD former or active smokers with at least a smoking history of 20 pack years
* Residual Volume (RV) >= 125% predicted value
* No Cardiac ultrasound signs of Cor Pulmonale

Exclusion Criteria:

* Acute Bronchial Exacerbation at recruitment
* Fertile women with age between 18 and 50 years old or with active period
* Pregnancy
* Subjects enrolled in other clinical trials or that have taken part in one of them in the month preceding the enrollment.
* FEV1/FVC more than 70% of predicted value in basal conditions
* FEV1 more than 70% of predicted value in basal conditions
* Residual Volume < 125% predicted value
* Known deficit of alpha 1 antitrypsin
* Subjects that underwent a Lung Volume Reduction Surgery (LVRS)
* Subjects with known positivity to Human Immunodeficiency Virus (HIV)
* Misuse of alcool or drugs
* Lack of compliance in performing respiratory tests
* Subjects not capable to follow the study prescriptions because of psychic disorders or language problems.
* Long Term Oxygen Therapy with flows > 6 litres per minute (l/min) at rest
* Cor Pulmonale
* Patients that cannot take Indacaterol for cardiologic reasons

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Effect of the decrease of residual volume and functional residual capacity on right cardiac performance assessing E/A and E/e' parameters on the mitral, pulmonary and tricuspid valve anulus, telediastolic pulmonary gradient, and venous pulmonary flow. | The assessment will be made at three different time points: 1) At baseline 2) sixty (60) minutes after indacaterol inhalation 3) a hundred eighty (180) minutes after indacaterol inhalation
  The right cardiac performance will be assessed throw trans-thoracic coor-doppler echocardiography. A trained technician will perform three echocardiographies at baseline, after 60 and 180 minutes after inhalation of indacaterol 150 mcg breezehaler. At every time point, after the echocardiographic assessment, a spirometric, plethysmographic and the lung diffusion for carbon monoxide test will be made in order to evaluate static and dynamic lung volumes.

SECONDARY OUTCOMES:
Evaluation of interventricular septum motility modification | The assessment will be made at three different time points: 1) At baseline 2) sixty (60) minutes after indacaterol inhalation 3) a hundred eighty (180) minutes after indacaterol inhalation
  Interventricular septum motility modifications will be assessed throw trans-thoracic coor-doppler echocardiography. A trained technician will perform three echocardiographies at baseline, after 60 and 180 minutes after inhalation of indacaterol 150 mcg breezehaler.
Evaluation of cardiac left ventricular ejection fraction modifications | The assessment will be made at three different time points: 1) At baseline 2) sixty (60) minutes after indacaterol inhalation 3) a hundred eighty (180) minutes after indacaterol inhalation
  Interventricular septum motility modifications will be assessed throw trans-thoracic coor-doppler echocardiography. A trained technician will perform three echocardiographies at baseline, after 60 and 180 minutes after inhalation of indacaterol 150 mcg breezehaler.
Evaluation of right cardiac chambers kinetics modifications | The assessment will be made at three different time points: 1) At baseline 2) sixty (60) minutes after indacaterol inhalation 3) a hundred eighty (180) minutes after indacaterol inhalation
  Interventricular septum motility modifications will be assessed throw trans-thoracic coor-doppler echocardiography. A trained technician will perform three echocardiographies at baseline, after 60 and 180 minutes after inhalation of indacaterol 150 mcg breezehaler.
Evaluation of inspiratory capacity modifications | A spirometric and plethysmographic assessment will be performed at three different time points: 1) At baseline 2) sixty (60) minutes after indacaterol inhalation 3) a hundred eighty (180) minutes after indacaterol inhalation
Evaluation of specific airway resistances modifications | A spirometric and plethysmographic assessment will be performed at three different time points: 1) At baseline 2) sixty (60) minutes after indacaterol inhalation 3) a hundred eighty (180) minutes after indacaterol inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Pierachille Santus, Md, PhD, Principal Investigator — Università degli Studi di Milano-Pneumologia Riabilitativa-Fondazione Salvatore Maugeri-MILANO
Locations (1):
- Pneumologia Riabilitativa-Fondazione Maugeri-Istituto Scientifico di Milano- IRCCS, Milan, Milan, Italy

REFERENCES:
- [Background] Steiropoulos P, Papanas N, Nena E, Bouros D. Indacaterol: a new long-acting beta2-agonist in the management of chronic obstructive pulmonary disease. Expert Opin Pharmacother. 2012 May;13(7):1015-29. doi: 10.1517/14656566.2012.674513. Epub 2012 Apr 4. PMID 22471750
- [Background] Barr RG, Bluemke DA, Ahmed FS, Carr JJ, Enright PL, Hoffman EA, Jiang R, Kawut SM, Kronmal RA, Lima JA, Shahar E, Smith LJ, Watson KE. Percent emphysema, airflow obstruction, and impaired left ventricular filling. N Engl J Med. 2010 Jan 21;362(3):217-27. doi: 10.1056/NEJMoa0808836. PMID 20089972